## The Effect of Interpersonal Relationships and Social Rhythm Therapy Individuals With Bipolar Disorder

The aim of this study was to determine the effectiveness of IPSRT based on Peplau's Interpersonal Relations theory, applied to individuals with bipolar disorder, on biological rhythm, interpersonal relationships and relapse frequency. It was planned as a follow-up study in a quantitative, randomized controlled experimental design. Pre-intervention pre-test, post-intervention post-test and follow-up scheme will be used.

This study is carried out with individuals with bipolar disorder registered in İzmir Katip Çelebi University Atatürk Training and Research Hospital Community Mental Health Center. Of the 60 patients enrolled here, 34 patients who met the research criteria and accepted the study were randomized to form the experimental and control groups. also "G. Using the "Power-3.1.9.2" program, the sample size at 80% confidence level was calculated before data collection. Accordingly, the effect size of the study was 0.40; (The minimum number of samples was calculated as 34 by taking the alpha value of 0.05 and the power of 0.80. In randomization, the patients were stratified by gender and Bipolar I - Bipolar II. After stratification, the participants were numbered, using the Research Randomizer site (https://www.randomizer.org/) individuals corresponding to the selected numbers were assigned to the experimental and control groups (experimental group: 17, control group: 17).

IPSRT based on Peplau Interpersonal Relations Theory will be applied to the experimental group. The control group will continue their follow-up and treatment at the Community Mental Health Center. Pre-test, post-intervention, post-intervention, 1st and 3rd month follow-ups were performed in both groups.

The data of the study were collected with Descriptive Information Form, Young Mania Rating Scale (YMÖ), Hamilton Depression Rating Scale (HAM-D), Biological Rhythm Evaluation Interview Form (BRDG), and Interpersonal Competence Scale - Short Form (BDS).

we cannot disclose the results as data collection is not yet complete